CLINICAL TRIAL: NCT05200520
Title: Improving Appetite Self-Regulation in Patients With Obesity: A Feasibility Study
Brief Title: Improving Appetite Regulation in Patients With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 21-2598
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Weight Loss; Weight Gain Prevention; Obesity
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Appetite Self-Regulation (Experimental): Participants will attend 12-weekly classes, delivered through virtual small group sessions (via zoom), self-monitor the participant's episodes of hunger and satiety with digital eating behavior website, weigh daily with a wireless Wi-Fi enabled scale, and use a FitBit to track physical activity. Participants will also receive weekly tailored feedback on eating, physical activity, and weight trends. Assessments will be conducted at 0, 3, and 6 months.
  Interventions: Behavioral: Appetite Self-Regulation Intervention

INTERVENTIONS:
Behavioral: Appetite Self-Regulation Intervention — The intervention will consist of content from Appetite Awareness Training (AAT), a cognitive-behavioral intervention to promote intuitive eating and the Diabetes Prevention Program (DPP)20, a behavioral lifestyle intervention. The goal of AAT is to enable participants to relearn their stomach's hunger signals and begin to obey and monitor functions of satiety. AAT has been successful in helping participants to reduce binge and overeating. Participants are taught to respond to external cues to eat (e.g., social gatherings), self-monitor the participant's adherence to biological signals of hunger and satiety, and to develop appropriate coping skills to manage urges to eat when not physically hungry.

SUMMARY:
Over 70% of U.S. adults have overweight or obesity. Currently, the most efficacious behavioral intervention for obesity is standard behavioral treatment (SBT), often composed of group sessions, calorie goals, and physical activity goals. With this approach, participants often lose 8-10% of the person's baseline weight, and also decrease risk for cardiovascular disease. Long-term weight loss, however, is limited; many participants return to baseline weight within five years following treatment. One reason SBT may not create long-term weight loss may be due to treatment components that teach participants to rely on external methods for changing eating decisions (e.g., counting calories, restricting certain foods), rather than internal cues of hunger and satiety. Because individuals with obesity report significant challenges with adhering to these cues, augmenting behavioral interventions with appetite self-regulation training may be a solution. Thus, the investigator propose to examine the feasibility and acceptability of a 6-month remotely-delivered appetite regulation + lifestyle modification intervention to treat obesity.

DETAILED DESCRIPTION:
Aim 1. Using a single-arm design, the investigator will examine the feasibility and acceptability of a 6-month, remotely-delivered, appetite self-regulation intervention for weight loss maintenance.

Aim 2. Examine the preliminary efficacy of the intervention on weight maintenance at 4 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age,
* BMI ≥ 25-45 kg/m^2,
* have and regularly use a smartphone,
* weight loss of 5% or more within the last 2 years
* complete the screening questionnaire

Exclusion Criteria:

* have no internet access,
* report a medical condition that could jeopardize the person's safety in a weight control program with diet and exercise guidelines
* are currently pregnant
* are in substance use treatment
* are involved in another weight reduction program
* have received prior or planned bariatric surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-03-05 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Feasibility (Recruitment): Total Number of Eligible Adults Enrolled in the Study | 3 Months
  Recruitment is defined as the number of potential eligible adults screened for the study versus the number of persons who enrolled in the study.
Feasibility (Retention): Percentage of Participants Retained in the Study | 3 months
  Percentage of eligible participants who were enrolled and retained in the study through the 6 months.
Feasibility (Retention): Percentage of Participants Retained in the Study | 6 months
  Percentage of eligible participants who were enrolled and retained in the study through the 6 months.
Feasibility (Attendance): Percentage of Intervention Sessions Attended | 3 months
  Percentage of intervention sessions attended for the duration of the study by each participant.

SECONDARY OUTCOMES:
Change in weight regain | 3 months
  Participant body weight will be measured by trained research staff using calibrated digital scales, with participants in light indoor clothing, with pockets emptied and belts and shoes removed.
Change in weight regain | 6 months
  Participant body weight will be measured by trained research staff using calibrated scales with participants in light indoor clothing, with pockets emptied and belts and shoes removed.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Goode, PhD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC-Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No